CLINICAL TRIAL: NCT01935999
Title: A Single Center Study to Assess the Safety and Performance of a One Piece Closed Pouch in Subjects With a Colostomy
Brief Title: One Piece Closed Pouch in Subjects With a Colostomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ConvaTec Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CC-0512-13-A741
Record Dates: First submitted 2013-07-29; First posted 2013-09-05 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-09

CONDITIONS: Colostomy
Keywords: Colostomy; peristomal skin; stoma; pouch

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- One piece closed pouch (Other): One piece closed pouch
  Interventions: Device: One piece closed pouch

INTERVENTIONS:
Device: One piece closed pouch — A one piece closed pouch for the collection of stool from a colostomy stoma
  Other Names: Enhanced one piece closed pouch

SUMMARY:
A study to assess the safety and performance of an enhanced one piece closed pouch in a 12 subjects with a colostomy.

DETAILED DESCRIPTION:
Twelve subjects are to be recruited into this 10 day single centre study to assess primarily safety in terms of adverse events and condition of the skin surrounding the stoma and condition of the stoma. Performance will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Of legal consenting age and able to provide written informed consent
* Is able to read, write, and understand the primary language of the investigative site.
* Have a colostomy for more than 3 months
* Currently a one or two piece closed or drainable pouch user (all attempts will be made to include ConvaTec Active Life or Esteem Plus one piece closed pouch users)
* Have unbroken peri-stomal skin (healthy normal skin to L1 on the SACs Instrument Scale # 1)
* Have a stoma considered 'normal' in appearance in accordance with the stoma, color, moisture and structure rating scales
* Be willing to wear a one piece closed pouch with moldable wafer according to the usual wear pattern of this type of pouch
* Be willing to participate in the trial for 10 days plus 1 visit prior to the in-residence study period.
* Be willing to remain in residence for 3 days at a central location
* Be willing to meet with the investigator for a total of nine scheduled visits.
* Be willing to discontinue the use of pastes, adhesive strips and rings/seals used to seal the area between the skin barrier wafer and stoma during the use of the study device
* Other than their colostomy considered to have a healthy/stable health status
* Have good manual dexterity and be able to take care of their stoma independently
* Be willing and able to complete a diary card for the duration of the study.
* Be willing to take photographs of the stoma and pouch on pouch removal

Exclusion Criteria:

* Subjects with a history of sensitivity to any one of the ostomy products or the components being studied
* Subjects with stoma duration of less than 3 months
* Subjects who currently use a belt with their usual appliance
* Subjects who have been entered into the study before, or who have previously taken part in a study in the last month.
* Subjects who require convexity or other skin fillers (pastes, seals, or rings) to even undulations of the peristomal skin
* Subjects undergoing chemotherapy or radiotherapy
* Subjects who have any other medical condition which, according to the investigator justifies exclusion from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Safety | 10 days - duration of study period
  Safety in relation to type and number of adverse events, condition of the skin surrounding the colostomy stoma and condition of the stoma

SECONDARY OUTCOMES:
Performance/Efficacy | 10 days duration of study period
  Performance/Efficacy of the pouch to stay in place and collect stool from the stoma. Ease of use, security will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Ann Popovich-Durnal, RN BSN, Principal Investigator — Unafilliated
Locations (1):
- Independent Nurse Consultants LLC, Tucson, Arizona, United States